CLINICAL TRIAL: NCT05000554
Title: The Safety and Efficacy of PD-1 Monoantrapical Chemotherapy in the Treatment of Local Advanced Stomach Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Quan Wang, Professor, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STARS-GC02
Record Dates: First submitted 2021-06-28; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Locally advanced gastric cancer (Experimental): Patients with locally advanced gastric cancer who can receive PD-1 monoclonal antibody combined with neoadjuvant chemotherapy
  Interventions: Procedure: Neoadjuvant Therapy

INTERVENTIONS:
Procedure: Neoadjuvant Therapy — Drug:
  Camrelizumab 200mg,d1，Repeat every 21 days for 3 courses； Oxaliplatin 130mg/m² ,d1;S-1 40-60mg,Bid, d1-14; S-1: bsa<1.25m2,40mg/time，twice a day；bsa1.25~1.5m2，50mg/time，twice a day；bsa≥1.5m2,60mg/次，twice a day，d1-d14；
  Procedure: Gastric cancer resection Distal gastrectomy combined with D2 lymph node dissection

SUMMARY:
To explore the safety and efficacy of local advanced stomach cancer patients receiving new complementary treatment of PD-1 monoantiotherapy before surgery

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven adenocarcinoma of the stomach, PD-L1+(CPS≥1).
2. Clinical cT3-4a/N+M0 disease, confirmed by upper gastrointestinal endoscopy and abdominal computed tomography (CT) and laparoscopy.
3. The gastric tumors are macroscopically resectable by distal gastrectomy with D2 lymph node dissection, and R0 or R1 resection can be achieved.
4. No bulky lymph node metastasis is detected by abdominal CT.
5. No pleural effusion, no ascites exceeding the pelvis and no metastasis to the peritoneum, liver or other distant organs are confirmed by abdominal pelvic CT.
6. No clinically apparent distant metastasis.
7. Karnofsky performance status ≥70%.
8. Sufficient oral intake.
9. No previous treatment with chemotherapy or radiation therapy for any tumors.
10. No previous surgery for the present disease.
11. Sufficient organ function, as evaluated by laboratory tests 7 days or more after the date when the anticancer drugs were given. When patients are recovering from myelosuppression,the revised criteria are shown in parentheses. White blood cell count≥3000/mm3 (2000/mm3) Platelet count≥10.0*104/mm3 (5.0*104/mm3) Aspartate aminotransferase≤100 IU/l Alanine aminotransferase≤100 IU/l Total bilirubin≤2.0 mg/dl Serum creatinine≤1.5 mg/dl
12. No need for emergency surgery due to bleeding or perforation of the primary tumor.
13. No mechanical obstruction.
14. Written informed consent.

Exclusion Criteria:

1. Past history of upper abdominal surgery.
2. Past history of surgery for the gastrointestinal tract.
3. Body mass index exceeding 30 kg/m2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 30 days
  Defined as the complete disappearance of tumor cells under a microscope after the completion of the neoadjuvant stomach cancer treatment.

SECONDARY OUTCOMES:
ORR | 30 days
  defined as the proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit. The sum of complete remission plus partial remission.
PFS | 3 years
  Defined as the time from the start of randomization to the progression of the disease or the death of the patient.
OS | 3 years
  Defined as the time between the beginning of randomization and the death of the patient for any reason.
postoperative complication | Up to 30 days post-operative
  Defined as postoperative complications that occur within 30 days of surgery, they are classified according to the Clavien-Dindo classification system.
operative mortality | Up to 30 days post-operative
  Defined as death of any cause within 30 days of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No